CLINICAL TRIAL: NCT03593746
Title: Effects of High Intensity Interval Training and Combined Training Associated With Photobiomodulation in Type 2 Diabetic (T2D) Patients: a Randomized Controlled Clinical Trial
Brief Title: Effects of High Intensity Interval Training and Combined Training in Type 2 Diabetic (T2D) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, LUCIANA MARIA MALOSA SAMPAIO, Professor of the postgraduate program in Rehabilitation Sciences, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T2Dexercise.photobiomodulation
Record Dates: First submitted 2018-05-07; First posted 2018-07-20 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; High-Intensity Interval Training; Exercise Training; Hyperglycaemia Due to Type 2 Diabetes Mellitus
Keywords: Cardiopulmonary Exercise Test; Rehabilitation; Diabetes Mellitus, Type 2; Functional Capacity; Photobiomodulation Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Physical Conditioning, Human; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT and LED therapy (Experimental): Light-Emitting Diode (LED) therapy followed by physical training with high intensity interval training (HIIT)
  Interventions: Other: Physical training; Other: Light-Emitting Diode (LED) therapy
- High intensity interval training (HIIT) (Sham Comparator): Light-Emitting Diode (LED) therapy simulation followed by physical training with high intensity interval training (HIIT)
  Interventions: Other: Physical training; Other: Light-Emitting Diode (LED) therapy
- Combined training and LED therapy (Experimental): Light-Emitting Diode (LED) therapy followed by physical training with combined training
  Interventions: Other: Physical training; Other: Light-Emitting Diode (LED) therapy
- Combined training (Sham Comparator): Light-Emitting Diode (LED) therapy simulation followed by physical training with combined training.
  Interventions: Other: Physical training; Other: Light-Emitting Diode (LED) therapy

INTERVENTIONS:
Other: Physical training — Type 2 diabetic patients will be subjected to different types of physical training (high intensity interval training or combined training).
Other: Light-Emitting Diode (LED) therapy — Type 2 diabetic patients will be subjected to Light-Emitting Diode (LED) therapy (active or sham).

SUMMARY:
Diabetes has become a widespread epidemic, primarily because of the increasing prevalence and incidence of type 2 diabetes (T2D). T2D is a significant cause of premature mortality and morbidity related to cardiovascular disease, blindness, kidney and nerve disease, and amputation.

Physical activity improves blood glucose control and can prevent or delay T2D, along with positively affecting lipids, blood pressure, cardiovascular events, mortality, and quality of life. At present, although physical activity is a key element in the prevention and management of T2D, the most effective exercise strategy (intensity, duration, and type of exercise) for improving glucose control and reducing cardiometabolic risk in type 2 diabetes has not been defined.

Studies with Light-Emitting Diode (LED) therapy have demonstrated its ability to promote pain relief, improve muscle and cardiopulmonary performance, minimize muscle fatigue, and stimulate wound healing. In relation to patients with T2D, who have prolonged conditions of hyperglycemia, studies to investigate the impact of photobiomodulation associated with physical training have not been found so far.

The objective of this study is to investigate the effects of different types of physical training associated with Light-Emitting Diode (LED) therapy on cardiometabolic status and quality of life in patients with T2D.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a significant health problem worldwide due to its high prevalence and mortality. It is chronic metabolic disorder characterized by hyperglycemia resulting from a relative deficiency in insulin through either reduced insulin secretion or reduced insulin action or both. The subsequent chronic hyperglycaemia causes glycation of tissues, which almost inevitably leads to acute disturbances in metabolism and long term end organ damage, especially the blood vessels, heart, and nerves, and severe health complications.

Individuals with T2D have reduced aerobic fitness characterized by lower peak pulmonary oxygen uptake. Many potential mechanisms could explain this impaired response, for example, reduced muscle blood flow and capillary density, defects in muscular oxygen diffusion, and lower mitochondrial oxygen utilization and function.

T2D is also associated with lower baroreflex sensitivity and abnormal chronotropic response, altering heart rate regulation. In addition, prolonged hyperglycemia in T2D causes a number of pathological changes in vascular endothelial cells, increasing the production of reactive oxygen species and inflammatory cytokines that cause mitochondrial dysfunction and oxidative damage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Confirmed diagnosis of type 2 diabetes;
* Sedentary lifestyle in the last six months, according to the criteria established by the American Heart Association (AHA).

Exclusion Criteria:

* Confirmed diagnosis of any (1) heart disease; (2) musculoskeletal disorder; (3) respiratory disease; (4) uncontrolled arterial hypertension; (5) peripheral neuropathy or (6) factors that limit the performance of any of the study evaluations and/or training.
* During the study, individuals with a presence of less than 80% in the training sessions will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | Change from Baseline to 12 weeks
  Oxygen consumption measurement during cardiopulmonary test
Incremental shuttle walking test | Change from Baseline to 12 weeks
  Distance in meters
Glycemic control | Change from Baseline to 12 weeks
  Evaluated by the percentage of glycated hemoglobin

SECONDARY OUTCOMES:
Autonomic Nervous System | Change from Baseline to 12 weeks
  Assesment by Heat Rate Variability analysis
Musculoskeletal Function | Change from Baseline to 12 weeks
  Muscular strength and endurance will be evaluated by Isokinetic Dynamometry
Physical Activity Questionnaire | Change from Baseline to 12 weeks
  The level of physical activity will be assessed using the international questionnaire short version physical activity (IPAQ). The continuous score allows assessing energy expenditure expressed in MET minutes/week. The IPAQ categories include: Insufficiently active (does not perform any physical activity); Sufficiently active (conducts vigorous activity at least three days a week >600 MET - 1400 MET); Very active (performs more than three days per week of vigorous activity 1500 MET - 3000 MET).
Endothelial Function | Change from Baseline to 12 weeks
  Endothelial function will be assessed by arterial flow-mediated dilation (FMD)
Quality of Life Questionary | Change from Baseline to 12 weeks
  Assesment by using the questionnaire Medical Outcomes Study 36 - Item Short - Form Health Survey (SF36). The SF-36 has eight sections (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning and Mental health). The scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability and higher scores = less disability.
Body mass index (BMI) | Change from Baseline to 12 weeks
  Weight and height will be combined to report BMI (kg/m2)
Other Biochemical Analyzes | Change from Baseline to 12 weeks
  Total cholesterol (Total-C) (mg/dl), low-density lipoprotein cholesterol (LDL-C) (mg/dl), high-density lipoprotein cholesterol (HDL-C) (mg/dl) and triglycerides (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana MM Sampaio, Professor, Principal Investigator — Nove de Julho University
Locations (1):
- UNINOVE, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bassi D, Mendes RG, Arakelian VM, Caruso FC, Cabiddu R, Junior JC, Arena R, Borghi-Silva A. Potential Effects on Cardiorespiratory and Metabolic Status After a Concurrent Strength and Endurance Training Program in Diabetes Patients - a Randomized Controlled Trial. Sports Med Open. 2016 Aug 11;2:31. doi: 10.1186/s40798-016-0052-1. eCollection 2015 Jun. PMID 27563535
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Karstoft K, Winding K, Knudsen SH, Nielsen JS, Thomsen C, Pedersen BK, Solomon TP. The effects of free-living interval-walking training on glycemic control, body composition, and physical fitness in type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2013 Feb;36(2):228-36. doi: 10.2337/dc12-0658. Epub 2012 Sep 21. PMID 23002086
- [Background] Chen L, Pei JH, Kuang J, Chen HM, Chen Z, Li ZW, Yang HZ. Effect of lifestyle intervention in patients with type 2 diabetes: a meta-analysis. Metabolism. 2015 Feb;64(2):338-47. doi: 10.1016/j.metabol.2014.10.018. Epub 2014 Oct 23. PMID 25467842
- [Background] Madsen SM, Thorup AC, Overgaard K, Jeppesen PB. High Intensity Interval Training Improves Glycaemic Control and Pancreatic beta Cell Function of Type 2 Diabetes Patients. PLoS One. 2015 Aug 10;10(8):e0133286. doi: 10.1371/journal.pone.0133286. eCollection 2015. PMID 26258597
- [Background] Francois ME, Little JP. Effectiveness and safety of high-intensity interval training in patients with type 2 diabetes. Diabetes Spectr. 2015 Jan;28(1):39-44. doi: 10.2337/diaspect.28.1.39. PMID 25717277
- [Background] Madsen SM, Thorup AC, Overgaard K, Bjerre M, Jeppesen PB. Functional and structural vascular adaptations following 8 weeks of low volume high intensity interval training in lower leg of type 2 diabetes patients and individuals at high risk of metabolic syndrome. Arch Physiol Biochem. 2015;121(5):178-86. doi: 10.3109/13813455.2015.1087033. Epub 2015 Oct 15. PMID 26471849
- [Background] Gibbs BB, Dobrosielski DA, Lima M, Bonekamp S, Stewart KJ, Clark JM. The association of arterial shear and flow-mediated dilation in diabetes. Vasc Med. 2011 Aug;16(4):267-74. doi: 10.1177/1358863X11411361. Epub 2011 Jun 27. PMID 21708874
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement executive summary. Diabetes Care. 2010 Dec;33(12):2692-6. doi: 10.2337/dc10-1548. No abstract available. PMID 21115771